CLINICAL TRIAL: NCT05306509
Title: Facilitating Early Integration of Palliative Care in Pediatric Oncology: Development and Implementation of a Nurse-initiated Conversation Program for Pediatric Cancer Patients and Their Families
Brief Title: Nurse-initiated Conversations for Early Integration of Palliative Care in Pediatric Oncology
Acronym: NiCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NiCE_21_427
Record Dates: First submitted 2022-03-20; First posted 2022-04-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor; Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-initiated conversations for early integration of palliative care (NiCE) (Experimental): Participants will receive nurse-initiated conversations facilitating early integration of palliative care in pediatric oncology.
  Interventions: Behavioral: NiCE
- Routine PPC (Other): Participants will be scheduled to meet with the PPC team only when participants themselves, their families, or the attending oncologist requested an appointment.
  Interventions: Other: Routine PPC

INTERVENTIONS:
Behavioral: NiCE — Participants will receive an initial conversation led by a trained senior nurse within eight weeks after initial oncologic diagnosis or relapse/recurrent disease diagnosis, with an introduction to the intervention and learning about the goals, values, hopes, and fears of each patient and family. The PPC team will then follow each patient by ongoing regular conversations (related to the child and family's conditions) led by the same nurse, every 4 weeks for six months, when symptom assessment and management, goal-directed supportive care, team collaboration, and care coordination will be delivered according to the family's needs. Increased PPC involvement, end-of-life care and bereavement care will be involved when necessary. If a participant feels any discomfort or distress during the intervention, a break will be taken until they feel better. If not, the central contact person will come and discussion about the participant's feeling and wiliness to continue the intervention.
  Arms: Nurse-initiated conversations for early integration of palliative care (NiCE)
Other: Routine PPC — Participants will be scheduled to meet with the PPC team only when participants themselves, their families, or the attending oncologist requested an appointment.
  Arms: Routine PPC

SUMMARY:
This study aims to develop and implement a pediatric palliative care (PPC) program. It is an open-label, randomized trial (2:1 randomization) in pediatric oncology department of Children's Hospital of Fudan University. The intervention group will receive Nurse-initiated Conversations for Early Integration of Palliative Care in Pediatric Oncology (NiCE). The control group will receive routine PPC (will be scheduled to meet with the PPC team only when participants themselves, their families, or the attending oncologist requested an appointment). The intervention will take 6 months.

DETAILED DESCRIPTION:
Early integration of PPC, endorsed by a number of international societies, is well supported by evidence on providing multi-layer relief in children and their families over the course of any life-threatening illness. This study will leverage oncology nurses' role, culturally adapt the well-recognized St. Jude Children's Individualized Care Planning and Coordination (ICPC) Model to develop and evaluate a nurse-initiated conversation program to facilitate early integration of palliative care in pediatric oncology care.

ELIGIBILITY:
Inclusion Criteria:

* Children within eight weeks of initial oncologic diagnosis or within eight weeks of relapse/recurrent disease diagnosis
* Children speaking Chinese
* Children's family caregivers accompanying the child in the hospital (only one family member is eligible to take this role under current hospital policy)
* Children's family caregivers speaking Chinese
* Health care providers who are taking care of the eligible children, including but not limited to physicians, nurses, and social workers

Exclusion Criteria:

- Children who, in the opinion of their physician, are not capable mentally or verbally of participating in the survey or interview

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Scores of children's quality of life | Measured every three months over six months.
  Scores of children's quality of life will be measured by Peds Quality of Life TM4.0 scale. It encompasses four subscales: physical, emotional, social and school functioning. It asks how much of a problem each item has been during the past month. It comprised of parallel child self-report and parent proxy-report formats. Child self-report includes ages 5-7 years (young child), ages 8-12 years (child), and ages 13-18 years (adolescent). All items use a five-point Likert response set range from 'never' to 'almost always'. Items are reverse-scored and linear-early transformed to a scale of 0 to 100 (0 = 100, 1= 75, 2= 50, 3= 25, 4=0), so that higher scores indicate a better quality of life. It is a repeated measurement, will be measured at baseline, three months and six months, for three times.

SECONDARY OUTCOMES:
Incidence of adverse events | Measured every four weeks over six months.
  Incidence of adverse events (AEs) will be measured by the Pediatric Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PED-PRO-CTCAE). This study will measure the incidence of 15 core AEs (abdominal pain, anorexia, nausea, vomiting, constipation, diarrhea, cough, pain, headache, neuropathy, mucositis, anxiety, depression, fatigue, insomnia), as perceived and reported by children 7 to 18 years of age or parent proxy (0-18 years), using a 7-day reference period with 4 response options per item. Presence of each of the 15 AEs will be measured as a dichotomous variable of the AE symptom (1-if any of the AEs happens; 0-none AEs). It is a repeated measurement, will be measured at baseline and every four weeks, for seven times.
Scores of children's mobility | Measured every three months over six months.
  Scores of children's mobility will be measured by Pediatric patient-reported outcomes measurement information system (Pediatric PROMIS) Short Form v2.0 - Mobility 8a. It can be reported by children 7 to 18 years of age or parent proxy (0-18 years) in relation to the past 7 days and in terms of a five-point response option range from 'never' to 'almost always' in most measures. Higher scores mean more of the measured symptom being experienced. The short form measure has 8 items and receives a T-score with a mean of 50 and a standard deviation of 10 based on the original reference sample. It is a repeated measurement, will be measured at baseline and every four weeks, for seven times.
Scores of children's family caregivers' care burden | Measured every three months over six months.
  Scores of children's family caregivers' care burden will be measured by Zarit Burden Inventory, by the family caregivers' self-reports. It is a 22-item, 5-point scale ranging from never (0) to always (4). A higher score indicates higher care burden. It is a repeated measurement, will be measured at baseline, three months and six months, for three times.
Scores of children's family caregivers' anxiety | Measured every three months over six months.
  Scores of children's family caregivers' anxiety will be measured by Zung's Self-Rating Anxiety Scale (SAS), by the family caregivers' self-reports. It is a 20-item, 4-point scale ranging from never (1) to often (4). The total score of 1.25 is the final standard score. A higher score indicates a severer anxiety symptom. It is a repeated measurement, will be measured at baseline, three months and six months, for three times.
Scores of children's family caregivers' depression | Measured every three months over six months.
  Scores of children's family caregivers' depression will be measured by Zung's Self-Rating Depression Scale (SDS) , by the family caregivers' self-reports. It is a 20-item, 4-point scale ranging from never (1) to often (4). The total score of 1.25 is the final standard score. A higher score indicates severer depressive symptoms. It is a repeated measurement, will be measured at baseline, three months and six months, for three times.
Acceptability of the NiCE intervention | At the sixth month of the study.
  Acceptability will be captured by interviews of family caregivers and healthcare workers about whether the content of this intervention is acceptable. Each participant will be asked about the same question: "Please tell me whether you think this intervention is acceptable? Please tell me more about your answer to this question". Acceptability will be defined when the participant clearly answered "yes".
Appropriateness of the NiCE intervention | At the sixth month of the study.
  Appropriateness will be assessed by interviews of family caregivers and healthcare workers of the intervention arm whether the content of this intervention is appropriate. Each participant will be asked about the same question: "Please tell me whether you think this intervention is appropriate? Please tell me more about your answer to this question". Appropriateness will be defined when the participant clearly answered "yes".
Feasibility of the NiCE intervention | At the sixth month of the study.
  Feasibility will be assessed by the number of nurses led conversations that actually occurred during the 6-month period.
Barriers and facilitators | At the sixth month of the study.
  Barriers and facilitators will be assessed by interviews of family caregivers and healthcare workers of the intervention arm. Each participant will be asked about the same two questions: (1) "Please tell me whether you think there is any barrier during the intervention? Please tell me more about your answer to this question". (2) "Please tell me whether you think there is any facilitators during the intervention? Please tell me more about your answer to this question".

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Zhai, MD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Hemotology/Oncology Unit and Surgical Oncology Unit of Children's Hospital of Fudan University, Shanghai, Minhang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt P, Otto M, Hechler T, Metzing S, Wolfe J, Zernikow B. Did increased availability of pediatric palliative care lead to improved palliative care outcomes in children with cancer? J Palliat Med. 2013 Sep;16(9):1034-9. doi: 10.1089/jpm.2013.0014. Epub 2013 Jul 31. PMID 23901834
- [Background] Snaman J, McCarthy S, Wiener L, Wolfe J. Pediatric Palliative Care in Oncology. J Clin Oncol. 2020 Mar 20;38(9):954-962. doi: 10.1200/JCO.18.02331. Epub 2020 Feb 5. PMID 32023163
- [Background] Haun MW, Estel S, Rucker G, Friederich HC, Villalobos M, Thomas M, Hartmann M. Early palliative care for adults with advanced cancer. Cochrane Database Syst Rev. 2017 Jun 12;6(6):CD011129. doi: 10.1002/14651858.CD011129.pub2. PMID 28603881
- [Background] Mahmood LA, Casey D, Dolan JG, Dozier AM, Korones DN. Feasibility of Early Palliative Care Consultation for Children With High-Risk Malignancies. Pediatr Blood Cancer. 2016 Aug;63(8):1419-22. doi: 10.1002/pbc.26024. Epub 2016 May 3. PMID 27148856
- [Background] Neuburg L. Early Initiation of Pediatric Palliative Care. J Pediatr Health Care. 2021 Jan-Feb;35(1):114-119. doi: 10.1016/j.pedhc.2020.05.006. Epub 2020 Jul 10. PMID 32660809
- [Background] Lafond DA, Kelly KP, Hinds PS, Sill A, Michael M. Establishing Feasibility of Early Palliative Care Consultation in Pediatric Hematopoietic Stem Cell Transplantation. J Pediatr Oncol Nurs. 2015 Sep-Oct;32(5):265-77. doi: 10.1177/1043454214563411. Epub 2015 Jan 23. PMID 25616372
- [Background] Levine DR, Johnson LM, Snyder A, Wiser RK, Gibson D, Kane JR, Baker JN. Integrating Palliative Care in Pediatric Oncology: Evidence for an Evolving Paradigm for Comprehensive Cancer Care. J Natl Compr Canc Netw. 2016 Jun;14(6):741-8. doi: 10.6004/jnccn.2016.0076. PMID 27283167
- [Background] Baker JN, Hinds PS, Spunt SL, Barfield RC, Allen C, Powell BC, Anderson LH, Kane JR. Integration of palliative care practices into the ongoing care of children with cancer: individualized care planning and coordination. Pediatr Clin North Am. 2008 Feb;55(1):223-50, xii. doi: 10.1016/j.pcl.2007.10.011. PMID 18242323